CLINICAL TRIAL: NCT05860023
Title: Effect of Pelvic Floor Muscle Strengthening and Aerobic Exercises on Uterus Involution
Brief Title: Exercises to Enhance Uterus Involution
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Omer Dursun, Asst. Prof., Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEUFTR-1
Record Dates: First submitted 2023-04-17; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Uterus Involution
Keywords: lactation; pregnancy; pelvic floor; pain
MeSH Terms: conditions — Breast Feeding; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Control group will take routine gynecologic treatment. Aerobic exercise group will attend to aerobic exercise programme for seven days. Aerobic exercise will be given with an intensity of 65% to 75% of the maximum heart rate of the individuals monitored by pulse oximeter.Aerobic exercise will take 30 minutes consisting of 5 minutes warm up, 20 minutes jogging, and 5 minutes cool down.
  Pelvic floor muscle strengthening group will be asked to perform six pelvic floor muscle strengthening exercise with moderate difficulty, recommended by the national association for incontinence for seven days. These exercises are straight leg raise, oblique reaches, partial curl up-obliques, pelvic tilt with crunch, quadruped hip extension, and bridge with adduction. Prior to discharge exercise sheet will be given to participants to do the exercises at home. Participants will be called daily to question their compliance to the exercise. Participants will be asked to keep exercise diary as well.
Who Masked: Outcomes Assessor
Masking Description: Interventions and assessment will be performed by separate researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): In this group, mothers will only take routine gynecologic. No additional treatment will be applied to the mothers in this group.
- Aerobic Exercise Group (Experimental): This group will attend to seven days aerobic exercise program with 65% to 75% of their maximum heart rate monitored with pulse oximeter. Aerobic exercise will take 30 minutes consisting of 5 minute warm up, 20 minute jogging and 5 minute cool down. Prior to discharge pulse oximeter will be given to the participants for self monitorization. Their compliance to exercise will be questioned with daily phone calls.
  Interventions: Other: Exercise
- Pelvic Floor Muscle Strengthening Group (Experimental): This group will attend to seven days pelvic floor muscle strengthening programme with moderate intensity consisting of 6 exercises recommended by the national association for incontinence. Prior to discharge exercise sheets will be given to the participants. Their compliance to exercise will be questioned with daily phone calls.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Individuals in the experimental group will be asked to perform aerobic exercise or pelvic floor muscle strengthening exercises.
  Arms: Aerobic Exercise Group; Pelvic Floor Muscle Strengthening Group

SUMMARY:
The goal of this randomized controlled study was to compare the effect of aerobic exercise and pelvic floor muscle strengthening exercises on uterus involution. In the scope of study following questions will be answered at the end of the study. First which of the exercise type is more effective to enhance uterus involution? Secondly, does exercises induce changes in lactation rate during the study period? Thirdly, does exercises improve the experienced pain? Study will be consisted of three groups as control group, pelvic floor exercise group and aerobic exercise group. Control group will take routine gynaecological treatment. Pelvic floor muscle strengthening exercise group will attend to seven day pelvic floor strengthening exercise programme. Aerobic exercise group will attend to seven day aerobic exercise programme consisting of walking.

DETAILED DESCRIPTION:
A total of 45 mothers who satisfies the eligibility criteria of the study will be recruited to the study. Following to the recruitment process mothers will be randomly assigned to the one of the three groups. Mothers in the control group will only take routine gynecologic treatment. Mothers in the aerobic exercise group will attend to aerobic exercises starting from the second day of the hospitalization for one week. Mothers who will be in pelvic floor strengthening exercise group after the randomization will be asked to perform six exercises with moderate difficulty that are recommended by the national association for incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Age of 19 to 35 years
* New born APGAR score is equal or higher than 8
* First pregnancy
* Giving birth in 37th to 40th weeks of the pregnancy
* Birthweight ranging from 2500 g to 4000 g

Exclusion Criteria:

* Eclampsia
* Puerperal psychosis
* Severe preeclampsia
* Multiple pregnancy story
* Uterus abnormality story
* Uterus surgery story
* Use of artificial estrogen
* Existence of systemic, mental or pregnancy related diseases
* Occurrence of complication during or after the pregnancy
* Symptoms of uterus subinvolution

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Mothers who gave birth to their first children will be recruited.
Enrollment: 45 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Uterus involution | Change from baseline uterus involution at one week
  To assess the uterus involution uterus volume, uterus diameters and thickness will be measured with ultrasound imaging. Ultrasound imaging will be performed in dorsal lithotomy position, without uterus activation, and with minimal uterus fullness. Uterus volume calculation will be performed with this formula: uterus anteroposterior diameter x uterus transverse diameter x uterus longitudinal diameter x 0.45.
Existence and Severity of Pain | Change from baseline pain at one week
  Pain will be assessed with visual analog scale (VAS). VAS consists of 10 cm horizontal line. At the one edge of the line 0 point is located meaning no pain, at the other edge 10 point is located meaning worst pain. Mothers will be asked to mark the point matching to their perceived pain. Minimal clinical significance of VAS is reported to be 1.1 or 1.2 cm.
  VAS and ultrasound imaging will be performed in first, second and eighth days of the study.

SECONDARY OUTCOMES:
Elapsed time from giving birth to first lactation | First day of the study
  Elapsed time will be recorded in minutes from giving birth to first lactation
Daily Lactation Time | Change from baseline daily lactation time at one week
  Daily lactation time and frequency will be calculated based on the mothers' reports.
Daily Lactation Frequency | Change from baseline daily lactation frequency at one week
  Daily lactation frequency will be calculated based on the mothers' reports.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Dursun, Asst. Prof., Principal Investigator — Bitlis Eren University; Burçhan Aydıner, M.D., Principal Investigator — Yuzuncu Yil University; Erhan Dincer, M.Sc., Principal Investigator — Bitlis Eren University; Özal Keleş, Ph.D., Principal Investigator — Bitlis Eren University; Yasemin Aslan Keleş, M.Sc., Principal Investigator — Biruni University
Locations (1):
- Van Yüzüncü Yıl University, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kristoschek JH, Moreira de Sa RA, Silva FCD, Vellarde GC. Ultrasonographic Evaluation of Uterine Involution in the Early Puerperium. Rev Bras Ginecol Obstet. 2017 Apr;39(4):149-154. doi: 10.1055/s-0037-1601418. Epub 2017 Apr 3. PMID 28371959
- [Background] Emshoff R, Bertram S, Emshoff I. Clinically important difference thresholds of the visual analog scale: a conceptual model for identifying meaningful intraindividual changes for pain intensity. Pain. 2011 Oct;152(10):2277-2282. doi: 10.1016/j.pain.2011.06.003. Epub 2011 Jul 2. PMID 21726939
- [Background] Tanaka H, Monahan KD, Seals DR. Age-predicted maximal heart rate revisited. J Am Coll Cardiol. 2001 Jan;37(1):153-6. doi: 10.1016/s0735-1097(00)01054-8. PMID 11153730
- [Background] Snyder AR, Greif SM, Clugston JR, FitzGerald DB, Yarrow JF, Babikian T, Giza CC, Thompson FJ, Bauer RM. The Effect of Aerobic Exercise on Concussion Recovery: A Pilot Clinical Trial. J Int Neuropsychol Soc. 2021 Sep;27(8):790-804. doi: 10.1017/S1355617721000886. PMID 34548116
- See also: Pelvic Floor Muscle Strengthening Exercises — https://nafc.org/downloadable-pelvic-floor-exercises/